CLINICAL TRIAL: NCT01856036
Title: CHUM-CRYOABLATION: Anti-Tumor Immunity Induced by Cryoablation of Invasive Breast Cancers
Brief Title: Anti-Tumor Immunity Induced by Cryoablation of Invasive Breast Cancers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institute and contacted IRB to close study.
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUM-CRYOABLATION
Record Dates: First submitted 2013-04-18; First posted 2013-05-17 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Ductal Histology; Unifocal; Estrogen Receptor Positive; her2neu negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoablation (Experimental): Cryoablation of breast cancer will be performed using a freeze-thaw technique and an IceCure probe. Cryoablation cycles will be determined by IceCure software programmed by the treating surgeon.
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — Cryoablation of breast cancer will be performed using a freeze-thaw technique and an IceCure probe. Cryoablation cycles will be determined by IceCure software programmed by the treating surgeon.

SUMMARY:
This protocol will study the impact of cryoablation on immune response in patients diagnosed with invasive breast cancers smaller than 1.5 cm. It will profile the immune response to cryoablation of invasive breast cancers. The intra-tumoral and systemic immune response to cryoablation will be determined and compared to pre-ablated breast cancer specimens and historical control specimens.

DETAILED DESCRIPTION:
Patients with small breast cancers will undergo cryoablation of their breast cancer. Approximately six weeks after cryoablation, definitive breast surgery will be performed. Blood will be drawn for research before cryoablation and surgery and at regular follow-up visits. Blood and tissue samples will be used to determine immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with an invasive breast cancer 1.5 cm or less
2. The breast cancer must be of ductal histology, unifocal, estrogen receptor positive and her2/neu negative.
3. The tumor must be visible by ultrasound and the subject must not have had prior surgical resection of the primary lesion.
4. A clip marking the breast cancer must have been placed at the time of initial diagnosis or will be placed prior to cryotherapy.
5. The breast cancer must be amenable to cryoablation (visible by ultrasound and more than 2 mm from skin or chest wall).
6. Subjects with metastatic disease at diagnosis who elect to have their primary tumor excised are eligible for enrollment.
7. For subjects with breast implants, the treating physician must document that adequate distance exists between the lesion and the implant to ensure that the ablated lesion with not contact or jeopardize the implant.
8. Subjects must be able to provide consent.

Exclusion Criteria:

1. Subjects with breast cancers of lobular histology, with lymph vascular invasion or extensive intraductal component will be excluded.
2. Subjects with multi-centric or multi-focal breast cancers
3. Subjects with breast cancers that have invaded skin or have significant skin tethering (assessed clinically).
4. Subjects receiving chemotherapy within one year or undergoing neoadjuvant chemotherapy are excluded.
5. Subjects with metastatic disease at diagnosis will be excluded unless they elect definitive surgical therapy for their primary lesion.
6. Subjects with breast cancers not amenable to cryoablation (lesions not visible by ultrasound, against the chest wall or within 2 mm of skin) will be excluded.
7. Subjects diagnosed with another malignancy in the preceding 5 years will be excluded.
8. Subjects diagnosed with simultaneous bilateral breast cancer.
9. Subjects receiving immunosuppressive therapy within 6 months including oral steroids will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Characterization of the intra-tumoral and systemic immune response to cryoablation in invasive breast cancers | 12 Months
  1. Determine number (percentage via flow cytometry), phenotype and functionality of tumor infiltrating lymphocytes in ablated breast cancer
  2. Determine number (percentage via flow cytometry)and phenotype of APC in ablated breast cancer
  3. Characterize cytokine and chemokine expression (in IU) in ablated tissue and in pre-ablated and post-ablated serum over time
  4. Quantify T cell response (IUs of IL2 and IFN gamma, and T cell specific cells as measured by number of spots on an elispot assay) to tumor associated antigens using in vitro assays of T cell proliferation and function (cytokine release, elispot, peptide-MHC)
  5. Determine morphology and histology of regional lymph node after cryoablation

SECONDARY OUTCOMES:
Comparison of the intra-tumoral and systemic response between non-ablated and ablated breast cancer and pre-ablated and post ablated serum | 24 Months
  1. Difference in intra-tumoral lymphocyte populations (percentage via flow cytometry) in ablated and non-ablated breast cancers
  2. Compare serum cytokine and chemokine expression (in IU) between patients undergoing or not undergoing tumor ablation
  3. Compare intra-tumoral lymphocyte populations (percentage via flow cytometry) in ablated tumor tissue with paraffin embedded specimens for tumors that are matched for age, tumor size and histology.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No